CLINICAL TRIAL: NCT02147678
Title: A Comparison Between Propofol and Etomidate in Hysteroscopy on Effect of Postoperative Sedation and Cognitive Function in Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wenying Song, Anesthesiologist, Shaanxi Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140522
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hysteroscopy; Hemodynamics; Sedation
MeSH Terms: interventions — Etomidate; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group E (Experimental): Etomidate/remifentanil group. Patients in group E will be given etomidate and remifentanil during the operation, the speeds are 10~15 μg/kg/min and 0.2~0.4 μg/kg/min, respectively.
  Interventions: Drug: Etomidate; Drug: Remifentanil; Drug: Anesthesia induction
- Group P (Experimental): Propofol/remifentanil group. Patients in group P will be given propofol and remifentanil during the operation, the speeds are 50~75 μg/kg/min and 0.2~0.4 μg/kg/min, respectively.
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Anesthesia induction

INTERVENTIONS:
Drug: Etomidate
  Other Names: Fu Er Li
  Arms: Group E
Drug: Propofol
  Arms: Group P
Drug: Remifentanil — During anesthesia maintenance, all patients will be given remifentanil at the speed of 0.2~0.4 μg/kg/min.
Drug: Anesthesia induction — For all patients, the induction protocol is midazolam 0.1 mg/kg, sufentanil 0.3 μg/kg, cisatracurium 0.15 mg/kg.

SUMMARY:
To compare the effect of propofol and etomidate in hysteroscopy on postoperative sedation and cognitive function in elderly patients

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 60 and 80 years
2. Selective hysteroscopic operation
3. American Society of Anesthesiology (ASA) Physical Status: Ⅰ or Ⅱ
4. Signed informed consent form
5. Expected operation duration is within 60 minutes

Exclusion Criteria:

1. Serious cardiac, cerebral, liver, kidney, lung, endocrine disease or sepsis
2. Long use of hormone or history of adrenal suppression
3. Allergy to trial drug or other contraindication
4. History or expected difficult airway
5. Identified, suspected abuse or long use of narcotic analgesia
6. Neuromuscular diseases
7. Mentally unstable or has a mental illness
8. Dysfunction of communication
9. Trend of malignant hyperthermia
10. Pregnant or breast-feeding women
11. Attended other trial past 30 days;

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Immediately after the entrance to the operating room until until 60 minutes after the operation
  heart rate will be recorded immediately after the entrance to the operating room, at the beginning of induction, 2.5 min, 5 min, 7.5 min, 10 min, 15 min, 20 min, 25 min and 30 min after the beginning of induction, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min and 60 min after the operation.
Mean arterial pressure | Immediately after the entrance to the operating room until until 60 minutes after the operation
  Mean arterial pressure will be recorded immediately after the entrance to the operating room, at the beginning of induction, 2.5 min, 5 min, 7.5 min, 10 min, 15 min, 20 min, 25 min and 30 min after the beginning of induction, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min and 60 min after the operation.
Pulse oxygen saturation | Immediately after the entrance to the operating room until until 60 minutes after the operation
  Pulse oxygen saturation will be recorded immediately after the entrance to the operating room, at the beginning of induction, 2.5 min, 5 min, 7.5 min, 10 min, 15 min, 20 min, 25 min and 30 min after the beginning of induction, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min and 60 min after the operation.
Respiratory rate | Immediately after the entrance to the operating room until until 60 minutes after the operation
  Respiratory rate will be recorded immediately after the entrance to the operating room, at the beginning of induction, 2.5 min, 5 min, 7.5 min, 10 min, 15 min, 20 min, 25 min and 30 min after the beginning of induction, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min and 60 min after the operation.
Narcotrend index | Immediately after the entrance to the operating room until until 60 minutes after the operation
  Narcotrend index will be recorded immediately after the entance to the operating room, at the beginning of induction, 2.5 min, 5 min, 7.5 min, 10 min, 15 min, 20 min, 25 min and 30 min after the beginning of induction, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min and 60 min after the operation.

SECONDARY OUTCOMES:
Cerebral injury parameters | Immediately after the entrance to the operating room until until 60 minutes after the operation
  2 ml blood will be collected immediately after the entrance to the operating room and 60 min after the operation, then SB-100 protein and neuron-specific enolase will be tested by enzyme-linked immunosorbent assay.
Length of stay | from the date of admission to the day of discharge, expected to 3 days
Score of Minimum Mental State Examination | 1 day before the operation to 45 minutes after the operation
  Score of Minimum Mental State Examination will be examined in preoperative visit, 10 minutes, 45 minutes after the operation
Verbal Fluency test | 1 day before the operation to 60 minutes after the operation
  Verbal Fluency test will be examined in preoperative visit and 60 minutes after the operation